CLINICAL TRIAL: NCT05491473
Title: Closed Incision Negative Pressure Therapy in Transverse Donor Site Closure of Free Profunda Artery Perforator Flap for Breast Reconstruction
Brief Title: Negative Pressure in PAP Donor Sites
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jung-Ju Huang, Associate Professor, Chang Gung Memorial Hospital
Other Study IDs: 202101649B0
Record Dates: First submitted 2022-08-03; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Breast Reconstruction
Keywords: breast reconstruction; profunda artery perforator flap; tensioned wound healing; negative pressure
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Patients who did not receive the application of iNPWT at the donor site.
- Negative pressure: Patients who received the application of iNPWT at the donor site.
  Interventions: Device: Closed incisional negative pressure wound therapy (iNPWT) system

INTERVENTIONS:
Device: Closed incisional negative pressure wound therapy (iNPWT) system — The closed incisional negative pressure wound therapy (iNPWT) system (PREVENA Incision Management System, KCI, an Acelity company, San Antonio, Texas, USA)
  Groups: Negative pressure

SUMMARY:
A retrospective chart review will be conducted to identify patients who received breast reconstruction using free profunda artery perforator (PAP) flap by the investigators from January 2015 to August 2021. The included patients will be grouped into two according to the application of incisional negative pressure wound therapy (NP) on the donor site. Patients' demographic data including their age at the surgery, body mass index (BMI), medical comorbidities including the hypertension and diabetes, and smoking history will be obtained from the retrospective chart review. Parameters of the flap will be carefully reviewed, including the flap harvested width, and flap harvested length, the flap harvested and used size, the size of the mastectomy, the ischemia time of the flap. The major interest is in the donor site management and patient's overall recovery. The complications of the donor site will be categorized into acute and chronic ones depending on the time of presence. Donor site complications, such as wound break down, hematoma, seroma, the total amount of the drainage will be recorded. The cutting time point for acute and chronic complications is 1 month. The total amount of drainage from the drainage tube inserted and the patients' off-bed time (day) will also be recorded. Besides, for patients with follow up time of more than 1 year, the scar will be evaluated using Vancouver scar scale.

Statistics Data will be analyzed using graphing and statistical analysis software SPSS 21 software (IBM, Chicago, Illinois, USA). Rank sum and independent t test will be applied to calculate continuous variables in demographic values, while Chi-square will be applied to calculate categorical variables such as postoperative complications. A probability of less than 0.05 will be considered significant.

Potential risks: No

Confidentiality:

All the patient identifiable information, which includes name, chart number and birthday, involved in the study will be strictly confidential.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent unilateral microsurgical breast reconstruction using PAP flaps from the PI (JJH) from November 2016 to August 2020

Exclusion Criteria:

* patients with delayed reconstruction

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received immediate breast reconstruction using PAP flaps by the PI from November 2016 to August 2020.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Off-bed time (days) | post-operative 14 days
Drainage amount (ml) | post-operative 14 days
Vacuum ball removed timing | post-operative 14 days
Vancouver Scar Scale (VSS) | 1 year after surgery
  Score range from 0-13, used to measure scar the scar appearance. The lower means a better outcome.
Re-open | post-operative 14 days
  Whether the patient return to the operation room to check the blood flow or re-do the anastomosis.
Donor site acute complication (< 30 days) | post-operative 30 days
Donor site chronic complication (> 30 days) | 1 year after surgery
Donor site revision | 1 year after surgery
  Whether the patient received scar revision surgery on the donor site where the tissue harvested for breast reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Ju Huang, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- ChangGungMH, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No